CLINICAL TRIAL: NCT03677596
Title: A PHASE 4, OPEN-LABEL, RANDOMIZED STUDY OF TWO INOTUZUMAB OZOGAMICIN DOSE LEVELS IN ADULT PATIENTS WITH RELAPSED OR REFRACTORY B-CELL ACUTE LYMPHOBLASTIC LEUKEMIA ELIGIBLE FOR HEMATOPOIETIC STEM CELL TRANSPLANTATION AND WHO HAVE RISK FACTOR(S) FOR VENO-OCCLUSIVE DISEASE
Brief Title: A Study Of Two Inotuzumab Ozogamicin Doses in Relapsed/ Refractory Acute Lymphoblastic Leukemia Transplant Eligible Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1931030; 2018-001557-27 (EudraCT Number)
Record Dates: First submitted 2018-07-27; First posted 2018-09-19 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-10

CONDITIONS: Leukemia; Precursor b-Cell Lymphoblastic Leukemia-Lymphoma; ACUTE LYMPHOBLASTIC LEUKEMIA
Keywords: Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; ACUTE LYMPHOBLASTIC leukemia; inotuzumab ozogamicin; Besponsa; transplant
MeSH Terms: conditions — Leukemia; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 2 phases: a run in phase and a randomized phase.
  Run in phase: a total of up to 22 patients will be enrolled to receive the starting dose of 1.2 mg/m2/cycle (dose level 2). A Simon Two Stage optimal design will be used. If acceptable efficacy (CR/CRi and MRD negativity) is observed in the run in phase, the study will enter the randomized phase.
  Randomized phase: if acceptable efficacy is observed in the run in phase, the study will enter the randomized phase. A total of approximately 80 patients will be randomized (1:1) to 1 of 2 dose levels of inotuzumab ozogamicin (40 patients per dose level).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dose Level 2 (Experimental): Inotuzumab ozogamicin at starting dose 1.2 mg/m2/cycle (administered in 3 divided doses). Most patients expected to receive 2 or 3 cycles (cycle length 21 to 28 days)
  Interventions: Drug: inotuzumab ozogamicin-dose level 2
- Dose Level 1 (Active Comparator): Inotuzumab ozogamicin at starting dose 1.8 mg/m2/cycle (administered in 3 divided doses). Most patients expected to receive 2 or 3 cycles (cycle length 21 to 28 days)
  Interventions: Drug: Inotuzumab ozogamicin-dose level 1

INTERVENTIONS:
Drug: inotuzumab ozogamicin-dose level 2 — Inotuzumab ozogamicin (BESPONSA™) is a CD22 targeted antibody drug conjugate (ADC) approved by US FDA for treatment of adults with relapsed or refractory B cell precursor acute lymphoblastic leukemia (ALL). The approved starting dose is 1.8mg/m2/cycle. This treatment arm evaluates a lower starting dose of 1.2mg/m2/cycle.
  Other Names: Besponsa
  Arms: Dose Level 2
Drug: Inotuzumab ozogamicin-dose level 1 — Inotuzumab ozogamicin (BESPONSA™) is a CD22 targeted antibody drug conjugate (ADC) approved by US FDA for treatment of adults with relapsed or refractory B cell precursor acute lymphoblastic leukemia (ALL). The approved starting dose of 1.8mg/m2/cycle is administered in this treatment arm.
  Other Names: Besponsa
  Arms: Dose Level 1

SUMMARY:
This study will explore 2 different doses of inotuzumab ozogamicin including the dose that is approved and a lower dose. The main purpose of this study is to evaluate whether a dose of inotuzumab ozogamicin, lower than the approved dose, could be recommended for adult patient with relapsed or refractory ALL who may be at higher risk for severe liver problems after inotuzumab ozogamicin treatment and stem cell transplant (a potentially curative therapy that can replace cancer cells with healthy cells). Efficacy and safety of the 2 doses will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory precursor CD22 positive B cell ALL with M2 or M3 marrow (≥5% blasts) and who are eligible for HSCT;
2. Have 1 or more of the following risk factors for developing VOD:

   1. Due to receive Salvage 2 or greater;
   2. Prior HSCT;
   3. Age ≥55 years.
   4. Ongoing or prior hepatic disease which may include a prior history of hepatitis or drug induced liver injury, as well as hepatic steatosis, nonalcoholic steatohepatitis, baseline elevations of bilirubin > upper limit of normal (ULN) and ≤1.5 x ULN.
3. Ph+ ALL patients must have failed treatment with at least 1 second or third generation tyrosine kinase inhibitor and standard multi agent induction chemotherapy;
4. Patients in Salvage 1 with late relapse should be deemed poor candidates for reinduction with initial therapy;
5. Patients with lymphoblastic lymphoma and bone marrow involvement 5% lymphoblasts by morphologic assessment;
6. Age 18 years to 75 years;
7. Eastern Cooperative Oncology Group (ECOG) performance status 0 2;
8. Adequate liver function, including total serum bilirubin ≤1.5 x ULN unless the patient has documented Gilbert syndrome, and aspartate and alanine aminotransferase (AST and ALT) ≤2.5 x ULN;
9. Serum creatinine ≤1.5 x ULN or any serum creatinine level associated with a measured or calculated creatinine clearance of >=40 mL/min;
10. Male and female patients of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for a minimum of 8 months (females) and 5 months (males) after the last dose of assigned treatment. A patient is of childbearing potential if, in the opinion of the Investigator, he/she is biologically capable of having children and is sexually active. Female subjects of nonchildbearing potential must meet at least 1 of the following criteria:

    1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state;
    2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
    3. Have medically confirmed ovarian failure. All other female subjects (including female subjects with tubal ligations) are considered to be of childbearing potential.
11. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study; patients with mental capacity which requires the presence of a legally authorized representative will be excluded from the study;
12. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Isolated extramedullary relapse (ie, testicular or central nervous system);
2. Burkitt's or mixed phenotype acute leukemia based on the WHO 2008 criteria;
3. Active central nervous system (CNS) leukemia, as defined by unequivocal morphologic evidence of lymphoblasts in the cerebrospinal fluid (CSF), use of CNS directed local treatment for active disease within the prior 28 days, symptomatic CNS leukemia (ie, cranial nerve palsies or other significant neurologic dysfunction) within 28 days. Prophylactic intrathecal medication is not a reason for exclusion;
4. Prior chemotherapy within 2 weeks before randomization with the following exceptions:

   1. To reduce the circulating lymphoblast count or palliation: ie, steroids, hydroxyurea or vincristine;
   2. For ALL maintenance: mercaptopurine, methotrexate, vincristine, thioguanine, and/or tyrosine kinase inhibitors.

   Patients must have recovered from acute non hematologic toxicity (to Grade 1 or less) of all previous therapy prior to enrollment.
5. Prior monoclonal antibodies within 6 weeks of randomization, with the exception of rituximab which must be discontinued at least 2 weeks prior to randomization;
6. Prior inotuzumab ozogamicin treatment or other anti CD22 immunotherapy within 6 months before randomization;
7. Prior allogeneic hematopoietic stem cell transplant (HSCT) within 90 days before randomization. Patients must have completed immunosuppression therapy for treatment of graft versus host disease (GvHD) prior to enrollment. At randomization, patients must not have Grade 2 or higher acute GvHD, or extensive chronic GvHD;
8. Peripheral absolute lymphoblast count >=10,000 /L (treatment with hydroxyurea and/or steroids/vincristine is permitted within 2 weeks of randomization to reduce the white blood cell [WBC] count);
9. Known systemic vasculitides (eg, Wegener's granulomatosis, polyarteritis nodosa, systemic lupus erythematosus), primary or secondary immunodeficiency (such as human immunodeficiency virus [HIV] infection or severe inflammatory disease);
10. Active hepatitis B infection as evidenced by hepatitis B surface antigen, active hepatitis C infection (must be anti-hepatitis C antibody negative or hepatitis C ribonucleic acid negative), or known seropositivity for HIV. HIV testing may need to be performed in accordance with local regulations or local practice;
11. Major surgery within 4 weeks before randomization;
12. Unstable or severe uncontrolled medical condition (eg, unstable cardiac function or unstable pulmonary condition);
13. Concurrent active malignancy other than non-melanoma skin cancer, carcinoma in situ of the cervix, or localized prostate cancer that has been definitely treated with radiation or surgery. Patients with previous malignancies are eligible provided that they have been disease free for >=2 years;
14. Patients with active heart disease or the presence of New York Heart Association (NYHA) stage III or IV congestive heart failure;
15. QTcF >470 msec (based on the average of 3 consecutive electrocardiogram [ECGs]);
16. Myocardial infarction within 6 months before randomization;
17. History of clinically significant ventricular arrhythmia, or unexplained syncope not believed to be vasovagal in nature, or chronic bradycardic states such as sinoatrial block or higher degrees of atrioventricular (AV) block unless a permanent pacemaker has been implanted;
18. Uncontrolled electrolyte disorders that can compound the effects of a QTc prolonging drug (eg, hypokalemia, hypocalcemia, hypomagnesemia);
19. Prior confirmed or ongoing hepatic veno occlusive disease (VOD) or sinusoidal obstruction syndrome (SOS), or other serious or current ongoing liver disease such as cirrhosis or nodular regenerative hyperplasia;
20. Administration of live vaccine within 6 weeks before randomization;
21. Evidence of uncontrolled current serious active infection (including sepsis, bacteremia, fungemia) or patients with a recent history (within 4 months) of deep tissue infections such as fascitis or osteomyelitis;
22. Patients who have had a severe allergic reaction or anaphylactic reaction to any humanized monoclonal antibodies;
23. Pregnant female subjects; breastfeeding female subjects; fertile male subjects and female subjects of childbearing potential who are unwilling or unable to use highly effective contraception as outlined in this protocol for the duration of the study and for a minimum of 8 months (females) and 5 months (males) after the last dose of investigational product;
24. Investigative site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study;
25. Participation in other studies involving investigational drug(s) within 2 weeks prior to study entry and/or during study participation (up through the end of treatment visit);
26. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2023-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- United States (7):
  - Keck Hospital of USC, Los Angeles, California
  - LAC+USC Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Rush University Medical Center, Chicago, Illinois
  - University of Maryland- Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Hungary (3):
  - Debreceni Egyetem Klinikai Központ, Orvosi Kepalkotó Klinika, Radiológia, Debrecen
  - Debreceni Egyetem Klinikai Központ, Pathológiai lntézet, Debrecen
  - Szabolcs-Szatmar Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Josa Andras Korhaz, Hematologia, Nyíregyháza
- India (6):
  - Artemis hospital, Gurugram, Haryana
  - Sahyadri Clinical Research and Development Centre, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital Nagar Road, Pune, Maharashtra
  - Christian Medical College, Vellore, Tamil Nadu
  - Christian Medical College Vellore- Ranipet Campus, Ranipet - 632517, Tamil Nadu, India
- Poland (4):
  - Klinika Hematologii i Transplantologii, Uniwersyteckie Centrum Kliniczne, Gdansk
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza - Radeckiego we Wroclawiu, Wroclaw
  - Apteka Centralna, Wroclaw
- Singapore (3):
  - National University Hospital, Singapore
  - Raffles Hospital, Singapore
  - Raffles Radiology, Singapore
- Spain (8):
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital General - Semisótano, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (2):
  - Changhua Christian Hospital, Changhua
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (11):
  - Anadolu Health Center Hospital, Gebze, Istanbul
  - Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital Clinical Research Center, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital Hematology Department, Ankara
  - Ankara University Faculty of Medicine Cebeci Hospital Hematology Department, Ankara
  - Private Medstar Antalya Hosp. Hematology and Stem Cell Transplantation Center, Antalya
  - Marmara University Pendik Training and Research Hospital Hematology Unit, Istanbul
  - Ege University Medical Faculty, Izmir
  - Dokuz Eylul University Medical Faculty, Izmir
  - Medicalpark Izmir Hospital, Izmir
  - Erciyes Universitesi Tip Fakultesi Hastaneleri, Kayseri
  - Ondokuz Mayis University Faculty Of Medicine Hospital, Samsun

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1931030

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 102 were enrolled. In Run-in Phase, 22 participants were enrolled and treated. In Randomized Phase, 80 participants were enrolled and treated.
Groups:
- 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized): Participants received a starting dose of inotuzumab ozogamicin 1.2 mg/m²/cycle (0.6 mg/m² on Day 1, 0.3 mg/m² on Days 8 and 15) intravenously. After complete remission (CR)/complete remission with incomplete hematologic recovery (CRi) is achieved, the dose was reduced to 0.9 mg/m²/cycle (0.3 mg/m² on Day 1, 8 and 15). The maximum treatment duration was approximately 52 weeks.
- 1.8 mg/m²/Cycle (Dose Level 1 Randomized Phase): Participants received a starting dose of inotuzumab ozogamicin 1.8 mg/m²/cycle administrated in 3 divided doses (0.8 mg/m² on Day 1, 0.5 mg/m² on Days 8 and 15) intravenously. After CR/CRi was achieved, the dose was reduced to 1.5 mg/m²/cycle (0.5 mg/m² on Days 1, 8 and 15) for 2-3 cycles. The cycle length was 21-28 days. The maximum treatment duration was approximately 52 weeks.
Period: Overall Study
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized Phase)
Started | 64 | 38
Completed | 41 | 19
Not Completed | 23 | 19
Not completed — Adverse Event | 0 | 1
Not completed — Death | 10 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Progressive Disease | 8 | 8
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Disease Relapse | 2 | 2
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who were randomized into the study.
Groups:
- 1.2 mg/m²/Cycle (Dose Level 2 Run-in): Participants received a starting dose of inotuzumab ozogamicin 1.2 mg/m²/cycle administrated in 3 divided doses (0.6 mg/m² on Day1, 0.3 mg/m² on Days 8 and 15) intravenously. After complete response (CR)/complete remission with incomplete hematologic recovery (CRi) was achieved, the dose was reduced to 0.9 mg/m²/cycle (0.3 mg/m² on Days 1, 8 and 15). The cycle length was 21-28 days. The maximum treatment duration was approximately 52 weeks.
- 1.2 mg/m²/Cycle (Dose Level 2 Randomized Phase): Participants received a starting dose of inotuzumab ozogamicin 1.2 mg/m²/cycle administrated in 3 divided doses (0.6 mg/m² on Day 1, 0.3 mg/m² on Days 8 and 15) intravenously. After CR/CRi was achieved, the dose was reduced to 0.9 mg/m²/cycle (0.3 mg/m² on Days 1, 8 and 15) for 2-3 cycles. The cycle length was 21-28 days. The maximum treatment duration was approximately 52 weeks.
- Total: Total of all reporting groups
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized Phase) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized Phase) | Total
Number analyzed (Participants) | 22 | 42 | 38 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 38 | 36 | 95
  >=65 years | 1 | 4 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 18 | 46
  Male | 12 | 24 | 20 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 3 | 10
  Not Hispanic or Latino | 20 | 36 | 35 | 91
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 6 | 11 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 17 | 34 | 25 | 76
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2 | 4
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is defined as: ECOG=0: Fully active, able to carry on all predisease performance without restriction; ECOG=1: Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, ie, light house work, office work; ECOG=2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    ECOG = 0 | 9 | 19 | 20 | 48
    ECOG = 1 | 13 | 20 | 13 | 46
    ECOG = 2 | 0 | 3 | 5 | 8
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] — BMI (kg/m^2) was computed as Height (cm)/Weight (kg) x 100.
  kg/m^2 | 24.98 [16 to 36] | 25.31 [17 to 39] | 24.78 [16 to 41] | 25.26 [16 to 41]
Body Surface Area (BSA) [Median (Full Range); unit: m^2] — BSA (m^2) will be computed using Du Bois Formula: 0.007184 x Weight (kg)^0.425 x Height (cm)^0.725.
  m^2 | 1.86 [1 to 2] | 1.82 [1 to 3] | 1.79 [1 to 3] | 1.80 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Veno-occlusive Disease (VOD)
Description: VOD happened when the small blood vessels that lead into the liver and were inside the liver become blocked. VOD is defined as: a. Classical VOD (first 21 days after HSCT): Bilirubin>=2 mg/dL and 2 (or more) of the following criteria must also be present: 1. Painful hepatomegaly; 2. Weight gain >5%; 3. Ascites. b. Late onset VOD (>21 days after HSCT): Classical VOD beyond Day 21; or Histologically proven VOD; or Two or more of the following criteria must be present: 1. Bilirubin >2 mg/dL; 2. Painful hepatomegaly; 3. Weight gain >5%; 4. Ascites. and hemodynamical and/or ultrasound evidence of VOD.
Time Frame: 2 years from randomization
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Groups:
- 1.2 mg/m²/Cycle (Dose Level 2 Randomized): Participants received a starting dose of inotuzumab ozogamicin 1.2 mg/m²/cycle (0.6 mg/m² on Day 1, 0.3 mg/m² on Day 8 and 15) intravenously. After CR/CRi is achieved, the dose was reduced to 0.9 mg/m²/cycle (0.3 mg/m² on Day 1, 8 and 15) for 2-3 cycles. The cycle length was 21-28 days. The maximum treatment duration was approximately 52 weeks.
- 1.8 mg/m²/Cycle (Dose Level 1 Randomized): Participants received a starting dose of inotuzumab ozogamicin 1.8 mg/m²/cycle (0.8 mg/m² on Day 1, 0.5 mg/m² on Day 8 and 15) intravenously. After CR/CRi is achieved, the dose was reduced to 1.5 mg/m²/cycle (0.5 mg/m² on Day 1, 8 and 15) for 2-3 cycles. The cycle length was 21-28 days. The maximum treatment duration was approximately 52 weeks.
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 22 | 42 | 64 | 38
Percentage of Participants | 9.1 | 14.3 | 12.5 | 5.3

2. Primary Outcome: Rate of Hematologic Remission (Complete Response [CR] / Complete Response With Incomplete Hematologic Recovery[CRi])
Description: CR is defined as a disappearance of leukemia as indicated by<5% marrow blasts and the absence of peripheral blood leukemic blasts, with recovery of hematopoiesis defined by absolute neutrophil count (ANC)>=1000/µL and platelets>=100000/µL. C1 extramedullary disease status is required. CRi is defined as CR except with ANC <1000/µL and/or platelets <100000/µL. C1 defined as complete disappearance of all measurable and non-measurable extramedullary disease with the exception of lesions with following must be true: For participants with>= 1 measurable lesion, all nodal masses>1.5cm in greatest transverse diameter (GTD) at baseline (last assessment before 1st dose of study treatment) must must have regressed to>=1.5cm in GTD and all nodal masses>=1cm & <=1.5cm in GTD at baseline have regressed to <1cm GTD or must have reduced by 75% in sum of products of greatest diameters. No new lesions. Spleen and other previously enlarged organs must have regressed in size and must not be palpable.
Time Frame: From first dose of study treatment of 6 cycles till follow-up up to 2 years, in total approximately 2.5 years
Population: All participants who were randomized into the study with study drug assignment based on randomization.
Measure: Number; unit: Percentage of Participants
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 22 | 42 | 64 | 38
Percentage of Participants | 50.0 | 83.3 | 71.9 | 68.4

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (All Causalities)
Description: Adverse event (AE) = any untoward medical occurrence in participant who received study treatment without regard to possibility of causal relationship. On-treatment period was defined as the period starting with the 1st dose of study treatment through 63 days after last dose or 1 day before start day of new anticancer therapy, whichever occurred first. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. All VOD cases were reported as SAE. Grades of severity were defined by Common terminology criteria for adverse events (CTCAE) v3.0. Grade 3=severe adverse event; Grade 4=life-threatening consequences; urgent intervention indicated. Grade 5=death related to AE. Results were reported as of the data cutoff date on 21 Sep 2022.
Time Frame: From first dose of study treatment drug through 63 days after last dose (approximately 52 weeks)
Population: All randomized participants who receive at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 22 | 42 | 64 | 38
Participants
  Participants with adverse events | 22 | 42 | 64 | 38
  Participants with SAEs | 15 | 28 | 43 | 21
  Participants with Maximum Grade 3 or 4 adverse events | 9 | 22 | 31 | 18
  Participants with Maximum Grade 5 adverse events | 7 | 11 | 18 | 10

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Treatment-related)
Description: Adverse event (AE) = any untoward medical occurrence in participant who received study treatment without regard to possibility of causal relationship. Treatment emergent AEs (TEAEs) were defined as AEs that reported the period starting with the first dose of study treatment drug through 63 days after last dose or 1 day before start day of new anticancer therapy, whichever occurred first. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Grades of severity were defined by CTCAE v3.0. Grade 3 = severe adverse event; Grade 4 = life-threatening consequences; urgent intervention indicated. Grade 5 = death related to AE. Causality of TEAEs were assessed by the Investigator. Results were reported as of the data cutoff date on 21 Sep 2022.
Time Frame: From first dose of study treatment drug through 63 days after last dose (approximately 52 weeks)
Population: All randomized participants who receive at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 22 | 42 | 64 | 38
Participants
  Participants with AEs | 13 | 18 | 31 | 22
  Participants with SAEs | 7 | 8 | 15 | 10
  Participants with Maximum Grade 3 or 4 AEs | 9 | 11 | 20 | 11
  Participants with Maximum Grade 5 AEs | 1 | 1 | 2 | 4

5. Secondary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (Post-HSCT)
Description: A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. All SAEs occurred after HSCT were reported in this OM. Results were reported as of the data cutoff date on 21 Sep 2022.
Time Frame: Starting from the first transplant after inotuzumab ozogamicin treatment and including the entire duration of subsequent follow up (approximately 52 weeks))
Population: All randomized participants who receive at least 1 dose of study drug and were post HSCT.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 10 | 21 | 31 | 12
Participants | 6 | 8 | 14 | 2

6. Secondary Outcome: Shift Summary of Hematology Laboratory Test Results From Grade <=2 at Baseline to Grade 3 or 4 Post-Baseline
Description: Baseline assessment was defined as the last assessment performed on or prior to the date of the first dose of study treatment. Following Parameters were analyzed for laboratory assessment: Hematology (Activated partial thromboplastin time prolonged, Anemia, Hemoglobin increased, International normalization rate (INR) increased, Leukocytosis, Lymphocyte count decreased, Lymphocyte count increased, Neutrophil count decreased, Platelet count decreased, White blood cell decreased). Grades of severity were defined by CTCAE v3.0. Grade 2 = moderate adverse event; Grade 3= severe adverse event; Grade 4 = life-threatening consequences; urgent intervention indicated. Results were reported as of the data cutoff date on 21 Sep 2022.
Time Frame: From first dose of study treatment drug through 63 days after last dose (approximately 52 weeks)
Population: All randomized participants who receive at least 1 dose of study drug and with at least 1 postbaseline assessment in each treatment group. 'Number analyzed' = Participants evaluable for this outcome measure for each specified row.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 22 | 42 | 64 | 38
Participants
  Activated partial thromboplastin time prolonged - Grade 3: number analyzed (Participants) | 19 | 31 | 50 | 27
  Activated partial thromboplastin time prolonged - Grade 3 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged - Grade 4: number analyzed (Participants) | 19 | 31 | 50 | 27
  Activated partial thromboplastin time prolonged - Grade 4 | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test.
  Anemia - Grade 3: number analyzed (Participants) | 15 | 22 | 37 | 20
  Anemia - Grade 3 | 8 | 13 | 21 | 11
  Anemia - Grade 4: number analyzed (Participants) | 15 | 22 | 37 | 20
  Anemia - Grade 4 | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test.
  Hemoglobin increased - Grade 3: number analyzed (Participants) | 6 | 12 | 18 | 13
  Hemoglobin increased - Grade 3 | 0 | 0 | 0 | 0
  Hemoglobin increased - Grade 4: number analyzed (Participants) | 6 | 12 | 18 | 13
  Hemoglobin increased - Grade 4 | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test.
  INR increased - Grade 3: number analyzed (Participants) | 11 | 16 | 27 | 12
  INR increased - Grade 3 | 0 | 0 | 0 | 0
  INR increased - Grade 4: number analyzed (Participants) | 11 | 16 | 27 | 12
  INR increased - Grade 4 | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test.
  Leukocytosis - Grade 3: number analyzed (Participants) | 7 | 11 | 18 | 13
  Leukocytosis - Grade 3 | 1 | 0 | 1 | 0
  Leukocytosis - Grade 4: number analyzed (Participants) | 7 | 11 | 18 | 13
  Leukocytosis - Grade 4 | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test.
  Lymphocyte count decreased - Grade 3: number analyzed (Participants) | 16 | 35 | 51 | 28
  Lymphocyte count decreased - Grade 3 | 1 | 15 | 16 | 7
  Lymphocyte count decreased - Grade 4: number analyzed (Participants) | 16 | 35 | 51 | 28
  Lymphocyte count decreased - Grade 4 | 4 | 2 | 6 | 4
  Lymphocyte count increased - Grade 3: number analyzed (Participants) | 13 | 14 | 27 | 17
  Lymphocyte count increased - Grade 3 | 2 | 1 | 3 | 3
  Lymphocyte count increased - Grade 4: number analyzed (Participants) | 13 | 14 | 27 | 17
  Lymphocyte count increased - Grade 4 | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test.
  Neutrophil count decreased - Grade 3: number analyzed (Participants) | 17 | 34 | 51 | 27
  Neutrophil count decreased - Grade 3 | 2 | 6 | 8 | 7
  Neutrophil count decreased - Grade 4: number analyzed (Participants) | 17 | 34 | 51 | 27
  Neutrophil count decreased - Grade 4 | 11 | 10 | 21 | 9
  Platelet count decreased - Grade 3: number analyzed (Participants) | 13 | 28 | 41 | 28
  Platelet count decreased - Grade 3 | 1 | 6 | 7 | 5
  Platelet count decreased - Grade 4: number analyzed (Participants) | 13 | 28 | 41 | 28
  Platelet count decreased - Grade 4 | 4 | 3 | 7 | 7
  White blood cell decreased - Grade 3: number analyzed (Participants) | 18 | 38 | 56 | 29
  White blood cell decreased - Grade 3 | 5 | 13 | 18 | 9
  White blood cell decreased - Grade 4: number analyzed (Participants) | 18 | 38 | 56 | 29
  White blood cell decreased - Grade 4 | 7 | 10 | 17 | 11

7. Secondary Outcome: Shift Summary of Chemistry Laboratory Test Results From Grade <=2 at Baseline to Grade 3 or 4 Post-Baseline
Description: Baseline assessment was defined as the last assessment performed on or prior to the date of the first dose of study treatment. Following Parameters were analyzed for laboratory assessment: Chemistry (Alanine aminotransferase increased, Alkaline phosphatase increased, Aspartate aminotransferase increased, Blood bilirubin increased, Chronic kidney disease, Creatinine increased, Gamma glutamyl transpeptidase (GGT) increased, Hypercalcemia, Hyperglycemia, Hyperkalemia, Hypermagnesemia, Hypernatremia, Hypoalbuminemia, Hypocalcemia, Hypoglycemia, Hypokalemia, Hypomagnesemia, Hyponatremia, Hypophosphatemia, Lipase increased and Serum amylase increased). Grades of severity were defined by CTCAE v3.0. Grade 2 = moderate adverse event; Grade 3= severe adverse event; Grade 4 = life-threatening consequences; urgent intervention indicated. Results were reported as of the data cutoff date on 21 Sep 2022.
Time Frame: From first dose of study treatment drug through 63 days after last dose (approximately 52 weeks)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- 1.2 mg/m²/Cycle (Dose Level 2 Run-in): Participants received a starting dose of inotuzumab ozogamicin 1.2 mg/m²/cycle administrated in 3 divided doses (0.6 mg/m² on Day1, 0.3 mg/m² on Days 8 and 15) intravenously. After complete response (CR)/complete remission with incomplete hematologic recovery (CRi) was achieved, the dose was reduced to 0.9 mg/m²/cycle (0.3 mg/m² on Days 1, 8 and 15). The cycle length was 21-28 days. The maximum treatment duration was approximately 52 weeks. The maximum treatment duration was approximately 52 weeks.
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 22 | 42 | 64 | 38
Participants
  Alanine aminotransferase increased - Grade 3: number analyzed (Participants) | 14 | 15 | 29 | 23
  Alanine aminotransferase increased - Grade 3 | 1 | 0 | 1 | 0
  Alanine aminotransferase increased - Grade 4: number analyzed (Participants) | 14 | 15 | 29 | 23
  Alanine aminotransferase increased - Grade 4 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased - Grade 3: number analyzed (Participants) | 14 | 28 | 42 | 22
  Alkaline phosphatase increased - Grade 3 | 1 | 0 | 1 | 1
  Alkaline phosphatase increased - Grade 4: number analyzed (Participants) | 14 | 28 | 42 | 22
  Alkaline phosphatase increased - Grade 4 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased - Grade 3: number analyzed (Participants) | 16 | 26 | 42 | 26
  Aspartate aminotransferase increased - Grade 3 | 1 | 3 | 4 | 0
  Aspartate aminotransferase increased - Grade 4: number analyzed (Participants) | 16 | 26 | 42 | 26
  Aspartate aminotransferase increased - Grade 4 | 0 | 0 | 0 | 0
  Blood bilirubin increased - Grade 3: number analyzed (Participants) | 14 | 17 | 31 | 20
  Blood bilirubin increased - Grade 3 | 1 | 1 | 2 | 0
  Blood bilirubin increased - Grade 4: number analyzed (Participants) | 14 | 17 | 31 | 20
  Blood bilirubin increased - Grade 4 | 0 | 0 | 0 | 0
  Chronic kidney disease - Grade 3: number analyzed (Participants) | 2 | 7 | 9 | 7
  Chronic kidney disease - Grade 3 | 0 | 0 | 0 | 0
  Chronic kidney disease - Grade 4: number analyzed (Participants) | 2 | 7 | 9 | 7
  Chronic kidney disease - Grade 4 | 0 | 0 | 0 | 0
  Creatinine increased - Grade 3: number analyzed (Participants) | 19 | 31 | 50 | 26
  Creatinine increased - Grade 3 | 0 | 0 | 0 | 0
  Creatinine increased - Grade 4: number analyzed (Participants) | 19 | 31 | 50 | 26
  Creatinine increased - Grade 4 | 0 | 0 | 0 | 0
  GGT increased - Grade 3: number analyzed (Participants) | 15 | 22 | 37 | 26
  GGT increased - Grade 3 | 1 | 2 | 3 | 3
  GGT increased - Grade 4: number analyzed (Participants) | 15 | 22 | 37 | 26
  GGT increased - Grade 4 | 0 | 0 | 0 | 0
  Hypercalcemia - Grade 3: number analyzed (Participants) | 10 | 12 | 22 | 15
  Hypercalcemia - Grade 3 | 0 | 0 | 0 | 0
  Hypercalcemia - Grade 4: number analyzed (Participants) | 10 | 12 | 22 | 15
  Hypercalcemia - Grade 4 | 0 | 0 | 0 | 0
  Hyperglycemia - Grade 3: number analyzed (Participants) | 13 | 24 | 37 | 21
  Hyperglycemia - Grade 3 | 2 | 2 | 4 | 2
  Hyperglycemia - Grade 4: number analyzed (Participants) | 13 | 24 | 37 | 21
  Hyperglycemia - Grade 4 | 0 | 0 | 0 | 0
  Hyperkalemia - Grade 3: number analyzed (Participants) | 10 | 11 | 21 | 14
  Hyperkalemia - Grade 3 | 0 | 0 | 0 | 0
  Hyperkalemia - Grade 4: number analyzed (Participants) | 10 | 11 | 21 | 14
  Hyperkalemia - Grade 4 | 1 | 0 | 1 | 0
  Hypermagnesemia - Grade 3: number analyzed (Participants) | 11 | 10 | 21 | 15
  Hypermagnesemia - Grade 3 | 1 | 0 | 1 | 1
  Hypermagnesemia - Grade 4: number analyzed (Participants) | 11 | 10 | 21 | 15
  Hypermagnesemia - Grade 4 | 0 | 0 | 0 | 0
  Hypernatremia - Grade 3: number analyzed (Participants) | 9 | 10 | 19 | 15
  Hypernatremia - Grade 3 | 0 | 0 | 0 | 0
  Hypernatremia - Grade 4: number analyzed (Participants) | 9 | 10 | 19 | 15
  Hypernatremia - Grade 4 | 0 | 1 | 1 | 0
  Hypoalbuminemia - Grade 3: number analyzed (Participants) | 16 | 15 | 31 | 21
  Hypoalbuminemia - Grade 3 | 1 | 3 | 4 | 3
  Hypoalbuminemia - Grade 4: number analyzed (Participants) | 16 | 15 | 31 | 21
  Hypoalbuminemia - Grade 4 | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test. | NA — Grade 4 was not applicable for this test.
  Hypocalcemia - Grade 3: number analyzed (Participants) | 12 | 16 | 28 | 15
  Hypocalcemia - Grade 3 | 1 | 0 | 1 | 0
  Hypocalcemia - Grade 4: number analyzed (Participants) | 12 | 16 | 28 | 15
  Hypocalcemia - Grade 4 | 0 | 0 | 0 | 0
  Hypoglycemia - Grade 3: number analyzed (Participants) | 10 | 12 | 22 | 16
  Hypoglycemia - Grade 3 | 0 | 0 | 0 | 0
  Hypoglycemia - Grade 4: number analyzed (Participants) | 10 | 12 | 22 | 16
  Hypoglycemia - Grade 4 | 0 | 0 | 0 | 0
  Hypokalemia - Grade 3: number analyzed (Participants) | 13 | 19 | 32 | 24
  Hypokalemia - Grade 3 | 1 | 2 | 3 | 1
  Hypokalemia - Grade 4: number analyzed (Participants) | 13 | 19 | 32 | 24
  Hypokalemia - Grade 4 | 1 | 0 | 1 | 0
  Hypomagnesemia - Grade 3: number analyzed (Participants) | 14 | 16 | 30 | 18
  Hypomagnesemia - Grade 3 | 1 | 0 | 1 | 1
  Hypomagnesemia - Grade 4: number analyzed (Participants) | 14 | 16 | 30 | 18
  Hypomagnesemia - Grade 4 | 0 | 0 | 0 | 1
  Hyponatremia - Grade 3: number analyzed (Participants) | 13 | 14 | 27 | 19
  Hyponatremia - Grade 3 | 1 | 0 | 1 | 0
  Hyponatremia - Grade 4: number analyzed (Participants) | 13 | 14 | 27 | 19
  Hyponatremia - Grade 4 | 0 | 0 | 0 | 0
  Hypophosphatemia- Grade 3: number analyzed (Participants) | 13 | 13 | 26 | 18
  Hypophosphatemia- Grade 3 | 2 | 0 | 2 | 1
  Hypophosphatemia - Grade 4: number analyzed (Participants) | 13 | 13 | 26 | 18
  Hypophosphatemia - Grade 4 | 0 | 0 | 0 | 1
  Lipase increased - Grade 3: number analyzed (Participants) | 15 | 23 | 38 | 24
  Lipase increased - Grade 3 | 3 | 3 | 6 | 2
  Lipase increased - Grade 4: number analyzed (Participants) | 15 | 23 | 38 | 24
  Lipase increased - Grade 4 | 0 | 2 | 2 | 0
  Serum amylase increased - Grade 3: number analyzed (Participants) | 14 | 18 | 32 | 22
  Serum amylase increased - Grade 3 | 1 | 1 | 2 | 0
  Serum amylase increased - Grade 4: number analyzed (Participants) | 14 | 18 | 32 | 22
  Serum amylase increased - Grade 4 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants Achieving a CR/CRi With Minimal Residual Disease (MRD) Negativity
Description: MRD was assessed by flow cytometry for CD22 and other cell surface markers associated with B-cell ALL. In participants who achieved CR/CRi, MRD negativity was defined as defined as <1 abnormal cell/10^4 nucleated cells by flow cytometry per central laboratory analysis.
Time Frame: At screening, once at Day 16-28 of Cycles 1 and 2, or until CR/CRi and MRD negativity were achieved, then after every 1-2 cycles as clinically indicated, and at EOT visit (maximum of 2.5 years)
Population: All participants who were randomized into the study and achieved CR/CRi.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 11 | 35 | 46 | 26
Participants | 8 | 25 | 33 | 18

9. Secondary Outcome: Duration of Remission (DoR) in Participants Achieving CR/CRi
Description: DoR was defined as time from date of first response in responders (CR/CRi) to the date of disease progression (i.e., objective progression, relapse from CR/CRi, including post-study treatment follow-up disease assessments) or death due to any cause, whichever occurs first. DoR was estimated using Kaplan-Meier methods. Results were reported as of the data cutoff date on 21 Sep 2022.
Time Frame: From first dose of study treatment of 6 cycles till follow-up up to 2 years, in total approximately 2.5 years
Population: Participants who were randomized into the study and with a remission (CR/CRi).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 11 | 35 | 46 | 26
Months | 5.2 [1.9 to NA] — The upper limit was not estimated due to fewer number of participants with event. | 6.5 [4.6 to 20.9] | 5.5 [4.6 to 20.9] | 6.8 [4.7 to 8.7]

10. Secondary Outcome: Progression-Free Survival
Description: PFS was defined as time from date of randomization to the date of disease progression (i.e., objective progression, relapse from CR/CRi, including post-study treatment follow-up disease assessments), death due to any cause, or starting new induction therapy/post-therapy HSCT without achieving CR/CRi, whichever occured first. PFS was estimated using Kaplan-Meier methods. Results were reported as of the data cutoff date on 21 Sep 2022.
Time Frame: From first dose of study treatment of 6 cycles till follow-up up to 2 years, in total approximately 2.5 years
Population: All participants who were randomized into the study with study drug assignment based on randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 22 | 42 | 64 | 38
Months | 2.9 [1.7 to 5.8] | 6.3 [4.8 to 10.0] | 5.3 [3.4 to 7.2] | 6.3 [2.8 to 8.0]

11. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from date of first dose of study treatment to death due to any cause. Participants without confirmation of death were censored at the date that the participant was last known to be alive. Results were reported as of the data cutoff date on 21 Sep 2022.
Time Frame: From first dose of study treatment of 6 cycles till follow-up up to 2 years, in total approximately 2.5 years
Population: All patients who were randomized into the study with study drug assignment based on randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 22 | 42 | 64 | 38
Months | 4.5 [3.2 to 8.6] | 9.6 [6.4 to NA] — The upper limit was not estimable due to fewer number of participants with event. | 7.6 [5.8 to 10.0] | 8.1 [5.4 to 10.4]

12. Secondary Outcome: Number of Participant Received HSCT Post Inotuzumab Ozogamicin Treatment
Description: Participants who underwent HSCT after inotuzumab ozogamicin treatment. Results were reported as of the data cutoff date on 21 Sep 2022.
Time Frame: From first dose of study treatment of 6 cycles till follow-up up to 2 years, in total approximately 2.5 years
Population: All participants who were randomized into the study with study drug assignment based on randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 22 | 42 | 64 | 38
Participants | 10 | 21 | 31 | 12

13. Secondary Outcome: The Cumulative Incidence Rate of Post-HSCT Relapse at Month 12
Description: Post-HSCT relapse is defined as the time from date of first HSCT after inotuzumab ozogamicin treatment to the date of first relapse post-HSCT. Cumulative incidence rates of an event at a particular timepoint were estimated with the CI calculated based on the cumulative incidence function using the method described by Kalbfleisch RL and Prentice JD. Results were reported as of the data cutoff date on 21 Sep 2022.
Time Frame: From first dose of study treatment to Month 12
Population: All participants who were randomized into the study with study drug assignment based on randomization and who were post HSCT.
Measure: Number (95% Confidence Interval); unit: Percentages of participants
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 10 | 21 | 31 | 12
Percentages of participants | 11.11 [0.40 to 41.66] | 22.53 [6.39 to 44.59] | 18.65 [6.46 to 35.72] | 16.67 [2.26 to 42.89]

14. Secondary Outcome: Number of Participants With Post-HSCT Mortality
Description: Post-HSCT Mortality was defined as the time from date of first HSCT after inotuzumab ozogamicin treatment to death due to any cause. Results were reported as of the data cutoff date on 21 Sep 2022.
Time Frame: From first dose of study treatment of 6 cycles till follow-up up to 2 years, in total approximately 2.5 years
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 10 | 21 | 31 | 12
Participants | 6 | 8 | 14 | 5

15. Secondary Outcome: Number of Participants With Post HSCT Non-Relapse Mortality
Description: Post HSCT non-relapse mortality was defined as time from date of first HSCT after inotuzumab ozogamicin treatment to death due to any cause without prior relapse. Results were reported as of the data cutoff date on 21 Sep 2022.
Time Frame: From first dose of study treatment of 6 cycles till follow-up up to 2 years, in total approximately 2.5 years
Population: All participants who were randomized into the study with study drug assignment based on randomization and who underwent HSCT after inotuzumab ozogamicin treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 10 | 21 | 31 | 12
Participants | 5 | 5 | 10 | 4

16. Secondary Outcome: Number of Participants With Post HSCT Relapse-Related Mortality
Description: Post HSCT Relapse-Related Mortality was defined as time from date of first HSCT after inotuzumab ozogamicin treatment to death due to any cause with prior relapse. Results were reported as of the data cutoff date on 21 Sep 2022.
Time Frame: From first dose of study treatment of 6 cycles till follow-up up to 2 years, in total approximately 2.5 years
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 10 | 21 | 31 | 12
Participants | 1 | 3 | 4 | 1

17. Secondary Outcome: Mean Predose Concentrations (Ctrough) of Inotuzumab Ozogamicin
Description: Ctrough was defined as the mean Predose concentration of study treatment.
Time Frame: Pre-dose on Cycle 1 Day 1, 8 and 15, and on Day1 and 8 of Cycle 2, 3 and 4.
Population: All treated participants who received at least 1 dose of study drug and had at least one PK sample collected and analyzed. 'Number analyzed' = Participants evaluable for this outcome measure for each specified row.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 22 | 42 | 64 | 38
ng/mL
  Cycle 1 Day 1 (C1D1): number analyzed (Participants) | 22 | 19 | 41 | 15
  Cycle 1 Day 1 (C1D1) | 1.9 (9.10) | 0.5 (1.97) | 1.3 (6.77) | 0.0 (0.00)
  C1D8: number analyzed (Participants) | 22 | 18 | 40 | 17
  C1D8 | 7.7 (20.53) | 5.0 (5.83) | 6.4 (15.61) | 5.4 (7.71)
  C1D15: number analyzed (Participants) | 21 | 18 | 39 | 12
  C1D15 | 8.9 (11.14) | 27.3 (52.32) | 17.4 (37.09) | 25.3 (19.47)
  C2D1: number analyzed (Participants) | 17 | 16 | 33 | 9
  C2D1 | 16.4 (21.43) | 18.8 (37.80) | 17.6 (30.02) | 39.7 (73.86)
  C2D8: number analyzed (Participants) | 18 | 17 | 35 | 10
  C2D8 | 42.6 (56.57) | 46.6 (50.89) | 44.6 (53.13) | 52.0 (27.94)
  C3D1: number analyzed (Participants) | 22 | 5 | 10 | 5
  C3D1 | 21.4 (18.46) | 13.2 (7.93) | 17.3 (14.09) | 27.5 (14.64)
  C3D8 | 31.9 (25.43) | 32.9 (12.96) | 32.5 (18.52) | 60.7 (44.89)
  C4D1: number analyzed (Participants) | 2 | 2 | 4 | 0
  C4D1 | 50.0 (14.64) | 25.5 (2.33) | 37.7 (16.53) |
  C4D8: number analyzed (Participants) | 2 | 3 | 5 | 1
  C4D8 | 48.7 (7.99) | 52.3 (9.56) | 50.8 (8.10) | 90.4 (NA) — Standard deviation was not applicable when there was only 1 participant analyzed.

18. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA)
Description: ADA incidence is defined as combined results of treatment-boosted and treatment-induced ADA-positive participants. The immunogenicity of inotuzumab ozogamicin was evaluated using a validated electrochemiluminescence (ECL)-based immunoassay.
Time Frame: At Day 1 of every cycle prior to the beginning of inotuzumab ozogamicin infusion and at the EOT visit, up to approximately 52 weeks.
Population: Participants who received at least 1 dose of study drug and had at least 1 ADA sample collected and analyzed for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 22 | 41 | 63 | 38
Participants
  Positive Predose ADA | 1 | 3 | 4 | 2
  Treatment-induced ADA | 1 | 0 | 1 | 1
  Treatment-boosted ADA | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Positive Neutralizing Antibody (NAb)
Description: NAb incidence is defined as combined results of treatment-boosted and treatment-induced NAb-positive participants. The immunogenicity of inotuzumab ozogamicin was evaluated using a validated electrochemiluminescence (ECL)-based immunoassay.
Time Frame: as for outcome 18
Population: Participants who received at least 1 dose of study drug and had at least 1 Nab sample collected and analyzed for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized)
Number analyzed (Participants) | 2 | 3 | 5 | 3
Participants
  Positive Predose NAb | 0 | 0 | 0 | 0
  Treatment-induced NAb | 0 | 0 | 0 | 0
  Treatment-boosted NAb | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment drug through 63 days after last dose or 1 day before start day of new anti-cancer therapy, whichever occurs first (approximately 52 weeks).
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety set. AEs were reported as of the data cutoff date on 21 Sep 2022.
Arm/Group | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized Phase) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized Phase)
All-Cause Mortality (participants affected / at risk) | 16/22 | 23/42 | 39/64 | 25/38
Serious Adverse Events (participants affected / at risk) | 15/22 | 28/42 | 43/64 | 21/38
Other Adverse Events (participants affected / at risk) | 18/22 | 32/42 | 50/64 | 29/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) (N=22) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized Phase) (N=42) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) (N=64) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized Phase) (N=38)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 4 | 7 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0
Coronary artery thrombosis (Cardiac disorders) | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Death (General disorders) | 0 | 1 | 1 | 1
Disease progression (General disorders) | 3 | 1 | 4 | 2
Pyrexia (General disorders) | 1 | 2 | 3 | 3
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 2 | 6 | 8 | 2
Graft versus host disease in liver (Immune system disorders) | 0 | 1 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 2 | 2 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 3 | 3 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 2 | 0 | 2 | 0
Fungal sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Hepatosplenic candidiasis (Infections and infestations) | 0 | 1 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 1 | 2 | 0
Sepsis (Infections and infestations) | 2 | 4 | 6 | 1
Septic shock (Infections and infestations) | 1 | 3 | 4 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Klebsiella test positive (Investigations) | 1 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 1 | 1 | 0
Focal dyscognitive seizures (Nervous system disorders) | 1 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 1 | 2
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in) (N=22) | 1.2 mg/m²/Cycle (Dose Level 2 Randomized Phase) (N=42) | 1.2 mg/m²/Cycle (Dose Level 2 Run-in + Randomized) (N=64) | 1.8 mg/m²/Cycle (Dose Level 1 Randomized Phase) (N=38)
Anaemia (Blood and lymphatic system disorders) | 2 | 9 | 11 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 3 | 4
Leukopenia (Blood and lymphatic system disorders) | 2 | 6 | 8 | 6
Neutropenia (Blood and lymphatic system disorders) | 4 | 16 | 20 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 14 | 19 | 13
Abdominal pain (Gastrointestinal disorders) | 2 | 5 | 7 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 3
Constipation (Gastrointestinal disorders) | 1 | 2 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 5 | 5 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 5 | 6 | 3
Asthenia (General disorders) | 0 | 1 | 1 | 2
Fatigue (General disorders) | 2 | 2 | 4 | 1
Pyrexia (General disorders) | 5 | 5 | 10 | 1
Influenza (Infections and infestations) | 2 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 4 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 2 | 2
Alanine aminotransferase increased (Investigations) | 5 | 5 | 10 | 3
Aspartate aminotransferase increased (Investigations) | 4 | 3 | 7 | 8
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 3 | 3
Blood lactate dehydrogenase increased (Investigations) | 2 | 3 | 5 | 4
Gamma-glutamyltransferase increased (Investigations) | 1 | 4 | 5 | 6
Neutrophil count decreased (Investigations) | 4 | 1 | 5 | 4
Platelet count decreased (Investigations) | 3 | 0 | 3 | 3
SARS-CoV-2 test positive (Investigations) | 0 | 2 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3 | 4 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Headache (Nervous system disorders) | 0 | 4 | 4 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2
Hypertension (Vascular disorders) | 2 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT03677596/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT03677596/SAP_001.pdf